CLINICAL TRIAL: NCT02698878
Title: Effects of Nutrition and Neuromuscular Electrical Stimulation on Local Glucose Uptake Into m. Soleus During 60 Days of Lower Leg Unloading
Brief Title: Unloading Induced Effects on Local Glucose Uptake Into m. Soleus
Acronym: NutriHEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DLR German Aerospace Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHP
Record Dates: First submitted 2016-02-23; First posted 2016-03-04 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Local Glucose Uptake; Glucose Metabolism Disorders
Keywords: Lupin Protein; Glucose Metabolism; GLUT4; Muscle Unloading; Neuromuscular Electrical Stimulation
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Control Group consisting of six healthy male subjects wearing only the HEPHAISTOS ORTHOSIS for lower leg unloading (60 days).
  Interventions: Device: HEPHAISTOS unloading orthotic device
- Intervention Group (Experimental): Intervention group consisting of seven healthy mal subjects, wearing the HEPHAISTOS orthosis for lower leg unloading (60 days), plus receiving lupin protein every day and performing a neuromuscular electrical stimulation training twice a day.
  Interventions: Dietary Supplement: lupin protein; Other: Neuromuscular electrical stimulation; Device: HEPHAISTOS unloading orthotic device

INTERVENTIONS:
Dietary Supplement: lupin protein — 19g of lupin crunchy every day for the whole duration of the intervention phase (60 days)
  Arms: Intervention Group
Other: Neuromuscular electrical stimulation — Individual neuromuscular electrical stimulation training had to be performed twice a day (morning and evening) over the whole duration of the intervention phase (60 days). Subjects were asked to continuously increase the intensity until a maximum intensity of 100mA per training.
  Other Names: NMES
  Arms: Intervention Group
Device: HEPHAISTOS unloading orthotic device — Orthotic device which unloads the muscles of the lower leg. Subjects had to wear the device for the whole duration of the intervention phase (60 days).
  Other Names: HEP

SUMMARY:
The present study aimed to investigate whether a daily intake of lupin protein and a neuromuscular electrical stimulation training twice a day can improve local glucose uptake into m. soleus during a 60 day unloading phase with a special unloading device, the HEPHAISTOS orthosis (HEP).

DETAILED DESCRIPTION:
The 60 day unloading intervention with the HEPHAISTOS unloading device had the following key objectives:

primary hypothesis:

* Assesment and evaluation of insulin sensitivity and local glucose uptake in the unloaded m. soleus and whether it can be improved by dietary supplementation of lupin seeds and neuromuscular electrical stimulation.

secondary hypotheses:

* Assesment and evaluation of unloading-induced reductions in muscle mass and whether they can be mitigated by dietary supplementation of lupin seed and neuromuscular electrical stimulation.
* Assesment and evaluation of whole-body glycemic effects of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers
* Age: between 20 and 45 years
* Body mass index (BMI): 20 -26 kg/m2
* Agreement and signed consent before the study

Exclusion Criteria:

* Smoker
* Competitive Athletes
* Diabetes mellitus
* Rheumatic disease
* Muscle or joint disease
* Bone fractures in the period up to one year before study start
* Herniated disc
* Flatfeet (pes planus)
* Allergy to nuts or legume
* Vascular diseases
* Epilepsy
* Severe hyperlipidemia
* Anemia (< Hb standard values; standard values healthy men: 13.5 -17.5 g/dl) *
* Increased thrombosis risk *
* Kidney disorder: deviations from normal values for creatinine in plasma. (Normal value: Creatinine < 1.20 mg/dl)*
* Lesions of the cruciate ligaments, or orthopedic surgery in the past 10 years on the side of the Hephaistos orthosis
* Achilles tendon injury, or rupture in the past 10 years on the side of the orthosis
* hyper-/hypocalcaemia (abnormal levels of calcium in the blood, normal level: 2.15 - 2.64 mmol/l)
* Intake of anti-inflammatory drugs during the study
* Abuse of drugs or alcohol (> than 20-30g alcohol/day)
* Participation in another clinical study within the last 2 months before the start of this study
* Increased bleeding tendency (hemophilia, regular use of anticoagulants)
* History of intolerance to local anesthetics
* Imprisoned during study
* Any other condition classed as unsuitable for study participation by the medical executive director
* prior convictions (objectionable criminal record)

Additional Exclusion Criteria for MRI

* Metal implants or other osteosynthesis material
* Pacemaker
* Claustrophobia

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in Local Glucose Uptake into m. soleus | Baseline to day 59 of the intervention phase
  Biopsies were taken from m. soleus
Changes in Local Glucose Metabolism in m. soleus | Baseline to day 60 of the intervention phase
  Microdialysis was performed in m. soleus

SECONDARY OUTCOMES:
Blood Glucose (changes in the whole body glucose metabolism) | Baseline and day 2 & 1 before the intervention phase, day 4, 14, 28, 42 & 60 of the intervention phase and day 2 & 14 after the intervention phase
Blood C-Peptide (changes in the whole body glucose metabolism) | Baseline and day 2 & 1 before the intervention phase, day 4, 14, 28, 42 & 60 of the intervention phase and day 2 & 14 after the intervention phase
Blood HbA1c (changes in the whole body glucose metabolism) | Baseline and day 2 & 1 before the intervention phase, day 4, 14, 28, 42 & 60 of the intervention phase and day 2 & 14 after the intervention phase
Blood Fructosamine (changes in the whole body glucose metabolism) | Baseline and day 2 & 1 before the intervention phase, day 4, 14, 28, 42 & 60 of the intervention phase and day 2 & 14 after the intervention phase
Insulin Sensitivity (changes in the whole body glucose metabolism) | Baseline and day 60 of the intervention phase
  Whole body insulin sensitivity assessed by hyperinsulinemic euglycemic clamp
Changes in Muscle Volume | Baseline to day 58 of the intervention phase
  Muscle volume measured by magnetic resonance imaging (MRI)
Changes in Muscle Function (jump performance) | Baseline to day 58 of the intervention phase
  A jump test was performed
Changes in Muscle Function (MVC) | Baseline to day 58 of the intervention phase
  Maximal voluntary contractions (MVC) - isometric and isokinetic - were performed
Compliance | During 60 days of intervention
  Electronic wearing time devices from Orthotimer were used to assess compliance of the subjects.
Movement | During 60 days of intervention and during 14 days of the recovery phase (post intervention phase)
  Accelerometers were used to assess movement of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jörn Rittweger, Prof. Dr., Study Director — DLR German Aerospace Center; Kathrin Schopen, M.Sc., Principal Investigator — DLR German Aerospace Center; Petra Frings-Meuthen, Dr., Principal Investigator — DLR German Aerospace Center

REFERENCES:
- [Derived] Zange J, Schopen K, Albracht K, Gerlach DA, Frings-Meuthen P, Maffiuletti NA, Bloch W, Rittweger J. Using the Hephaistos orthotic device to study countermeasure effectiveness of neuromuscular electrical stimulation and dietary lupin protein supplementation, a randomised controlled trial. PLoS One. 2017 Feb 16;12(2):e0171562. doi: 10.1371/journal.pone.0171562. eCollection 2017. PMID 28207840